CLINICAL TRIAL: NCT06391957
Title: Spirulina Supplementation In Recovery From Damaging Exercise
Acronym: SPIRAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4530276
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Damage Muscle
Keywords: spirulina; exercise recovery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina supplement (Experimental): 3g of spirulina supplement three times daily for 5 days.
  Interventions: Dietary Supplement: Spirulina supplement; Procedure: Eccentric exercise
- Placebo supplement (Placebo Comparator): macronutrient matched placebo supplement three times daily for 5 days.
  Interventions: Procedure: Eccentric exercise; Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Spirulina supplement — Participants consume a 3g spirulina supplement 3 times daily for 5 consecutive days.
  Arms: Spirulina supplement
Procedure: Eccentric exercise — On the morning of Day 3 (where Day 1 is when participants start taking supplements), participants perform a single bout of eccentric exercise. The exercise protocol is performed on a single leg and involves 300 (10 sets of 30 repetitions separated by 120 seconds) voluntary maximal, isokinetic, eccentric contractions of the knee extensor. Exercise is performed using a Biodex System 3 isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, USA), and contractions are performed at 60◦/s over an 80◦ range of motion.
Dietary Supplement: Placebo supplement — Participants consume a macronutrient matched placebo supplement 3 times daily for 5 consecutive days.
  Arms: Placebo supplement

SUMMARY:
Exercise can cause muscle damage, leading to a loss in muscle function, increased muscle soreness and inflammation. Evidence supports the use of nutritional strategies to help recovery. Spirulina is a type of algae. It is eaten as a food supplement as it is full of micronutrients, some which provide anti-inflammatory benefits. This work will assess the impact of taking spirulina supplements on recovery from hard exercise. Investigators will measure changes in muscle function, soreness and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Are available and willing to attend St Luke's Campus, Exeter
* Age 18 - 40
* BMI 18.5 - 30 kg/m2
* The participant exercises / plays sport for > 2 h/week, but doesn't do structured resistance strength training
* Self-reported as healthy (absence of injury or disease)
* Have no known food allergy to algae
* Are not taking any over the counter or prescribed medication that might interfere with study, e.g. anti-inflammatory medication
* Non-smoker

Exclusion Criteria:

* Are unable to attend St Luke's Campus, Exeter
* Are out-with age range 18 - 40
* BMI below 18.5 or above 30 kg/m2
* The participant does not exercise
* The participant does regular structured resistance strength training
* Known injury or disease that might influence study outcomes
* Have a known food allergy to algae
* Are taking over the counter or prescribed medication that might interfere with study, e.g. anti-inflammatory medication
* Smoker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Measure changes in the concentration of blood plasma inflammatory markers via immunoassay. | Measurements take place across a 6 day experimental period.
  Blood plasma inflammatory markers will be measured before (baseline) and after eccentric exercise (at 3, 6, 24, 48 and 72 h post eccentric exercise) in both the spirulina and placebo group. Inflammatory markers that will be assessed include: interferon γ (IFN-γ), interleukin (IL) -1β, -4, -6, -10, tumour necrosis factor α (TNF-α) via immunoassay (pg/mL).

SECONDARY OUTCOMES:
Measure changes in muscle function of the quadriceps using knee extensor peak isometric torque on a Biodex System 3 isokinetic dynamometer. | Measurements take place across a 6 day experimental period.
  Knee extensor peak isometric torque (three maximal isometric contractions at 75◦ of knee flexion) will be measured before (baseline) and after eccentric exercise (at 3, 6, 24, 48 and 72 h post eccentric exercise) in both the spirulina and placebo group to report recovery of peak isometric torque (N). Testing will be performed on a Biodex System 3 isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, US).
Measure changes in muscle function of the quadriceps using knee extensor total isokinetic work on a Biodex System 3 isokinetic dynamometer. | Measurements take place across a 6 day experimental period.
  Knee extensor total isokinetic work (area under the torque-time curve after 30 maximal, concentric, isokinetic knee extensor contractions performed at 75◦/s through an 80◦ range of motion) will be measured before (baseline) and after eccentric exercise (at 3, 6, 24, 48 and 72 h post eccentric exercise) in both the spirulina and placebo group to report recovery of total isokinetic work (N.s). Testing will be performed on a Biodex System 3 isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, US).
Measure changes in perceived lower body muscle soreness via visual analogue scale questionnaire. | Measurements take place across a 6 day experimental period.
  Perceived lower body muscle soreness will be measured before (baseline) and after eccentric exercise (at 3, 6, 24, 48 and 72 h post eccentric exercise) in both the spirulina and placebo group to report recovery of muscle. Participants will stand from a seated position and rate the corresponding sensation of lower body muscle soreness on a 100-mm visual analogue scale anchored by 'no pain' at 0 mm and 'worst possible pain' at 100 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, United Kingdom